CLINICAL TRIAL: NCT00990262
Title: Accuracy of Contrast Enhanced Multidetector Computed Tomography to Identify Cardiac Cause of Symptoms in Patients With Intermediate Likelihood of Acute Coronary Syndrome (ACS) - A Comparison to Standard Care
Brief Title: Rule Out Myocardial Infarction by Computer Assisted Tomography
Acronym: ROMICAT
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Udo Hoffmann, MD MPH, Massachusetts General Hospital
Other Study IDs: 2003P000458; R01HL080053-01 (NIH)
Record Dates: First submitted 2009-09-30; First posted 2009-10-06 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Unstable Angina Pectoris
Keywords: acute chest pain; emergency department; cardiac computed tomography
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Angina, Unstable; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute Chest Pain: Patients who presented to the emergency department with acute chest pain, with negative initial biomarkers and normal or non-ischemic ECG
  Interventions: Radiation: Cardiac Computed Tomography

INTERVENTIONS:
Radiation: Cardiac Computed Tomography — 1. Localization of the heart position in a projectional topographic scan of the chest.
  2. Determination of contrast agent transit time: 10 ml contrast agent.
  3. CT coronary angiography: CT scan in spiral acquisition mode with 330 ms rotation time, 32 x 0.6 mm collimation, a pitch of 2.8 mm/rotation, tube voltage of 120 kVp, and maximum tube current of 850 mA. 80 ml of contrast agent, followed by 40 ml saline solution will be injected at a rate of 4 ml/s. The mean breath hold duration for this acquisition is approximately 13 seconds.

SUMMARY:
The goal of this research is to determine noninvasively whether detection of coronary stenosis and plaque by multidetector computed tomography (MDCT) in patients with acute chest pain suspected of acute coronary syndrome (ACS) enhances triage, reduces cost and is cost effective. Among the 5.6 million patients with ACP presenting annually in emergency departments (ED) in the United States, a subgroup of two million patients is hospitalized despite normal initial cardiac biomarker tests and electrocardiogram (ECG). This subgroup is at low (20%) risk for ACS during the index hospitalization. Most (80-94%) patients with a diagnosis of ACS have a significant epicardial coronary artery stenosis ( >50% luminal narrowing). However, in -10% of patients non-stenotic coronary plaque triggers events, i.e. vasospasms, leading to myocardial ischemia. Since the absence of plaque excludes a coronary cause of chest pain, these patients could in theory be discharged earlier reducing unnecessary hospital admissions. Recent publications demonstrate high sensitivity and specificity of MDCT for the detection of significant coronary stenosis compared with coronary angiography and the detection of coronary plaque as validated with intravascular ultrasound. Using 64- slice MDCT we propose to study 400 patients with ACP, negative initial cardiac biomarkers and non-diagnostic ECG. We will analyze MDCT images for the presence of significant coronary artery stenosis and plaque and correlate the data with the clinical diagnosis of ACS (AHA guidelines) during the index hospitalization to determine the sensitivity and specificity. MDCT data, risk factors, and the results of standard diagnostic tests available at the time of MDCT will be used to generate a multivariate prediction function and derive a clinical decision rule. Based on this decision rule we will compare the diagnostic accuracies and cost effectiveness of competing strategies. We hypothesize that an MDCT- based diagnostic strategy will reduce the time to diagnosis of ACS, number of hospitalizations, and absolute cost of management of patients with acute chest pain compared to standard clinical care and is cost effective.

ELIGIBILITY:
Inclusion Criteria:

* Patients with any episode > five minutes of chest pain being admitted to rule out acute coronary syndrome

Exclusion Criteria:

* Positive initial troponin or CK-MB tests
* Diagnostic ECG changes (ST- segment elevation or horizontal ST- segment depression in more than two contiguous leads)
* Unstable clinical condition (hemodynamically unstable, ventricular tachycardia, persistent chest pain despite adequate therapy)
* Creatinine Clearance <50 mL/min
* Known allergy to iodinated contrast agents
* Patients on metformin therapy unable or unwilling to discontinue therapy for 48 hours after CT scan procedure
* Known asthma, reactive airway disease
* Patients currently in atrial fibrillation
* Previous intolerance to beta blocker
* Patients that are referred for coronary angiography/PCI by their PCP or cardiologist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who presented to the emergency department at Massachusetts General Hospital, with acute chest pain and with initial negative biomarkers and normal or non-ischemic ECG
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2005-05; Primary Completion 2007-05 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Accuracy of CT derived features of coronary artery disease and LV function for ACS | ED presentation to hospital discharge

SECONDARY OUTCOMES:
Major adverse cardiac events (MACE) - defined as death, myocardial infarction or coronary revascularization | Follow up at 6 months and 2 year after index hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Udo Hoffmann, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Truong QA, Bamberg F, Mahabadi AA, Toepker M, Lee H, Rogers IS, Seneviratne SK, Schlett CL, Brady TJ, Nagurney JT, Hoffmann U. Left atrial volume and index by multi-detector computed tomography: comprehensive analysis from predictors of enlargement to predictive value for acute coronary syndrome (ROMICAT study). Int J Cardiol. 2011 Jan 21;146(2):171-6. doi: 10.1016/j.ijcard.2009.06.029. Epub 2009 Jul 16. PMID 19615769
- [Background] Manini AF, Dannemann N, Brown DF, Butler J, Bamberg F, Nagurney JT, Nichols JH, Hoffmann U; Rule-Out Myocardial Infarction using Coronary Artery Tomography (ROMICAT) Study Investigators. Limitations of risk score models in patients with acute chest pain. Am J Emerg Med. 2009 Jan;27(1):43-48. doi: 10.1016/j.ajem.2008.01.022. PMID 19041532
- [Background] Lehman SJ, Schlett CL, Bamberg F, Nieman K, Abbara S, Hoffmann U. Appearance of acute and chronic coronary occlusions in contrast-enhanced cardiac computed tomography. JACC Cardiovasc Imaging. 2008 Nov;1(6):809-11. doi: 10.1016/j.jcmg.2008.07.016. Epub 2008 Nov 18. No abstract available. PMID 19356518
- [Result] Hoffmann U, Bamberg F, Chae CU, Nichols JH, Rogers IS, Seneviratne SK, Truong QA, Cury RC, Abbara S, Shapiro MD, Moloo J, Butler J, Ferencik M, Lee H, Jang IK, Parry BA, Brown DF, Udelson JE, Achenbach S, Brady TJ, Nagurney JT. Coronary computed tomography angiography for early triage of patients with acute chest pain: the ROMICAT (Rule Out Myocardial Infarction using Computer Assisted Tomography) trial. J Am Coll Cardiol. 2009 May 5;53(18):1642-50. doi: 10.1016/j.jacc.2009.01.052. PMID 19406338
- [Result] Mahabadi AA, Bamberg F, Toepker M, Schlett CL, Rogers IS, Nagurney JT, Brady TJ, Hoffmann U, Truong QA. Association of aortic valve calcification to the presence, extent, and composition of coronary artery plaque burden: from the Rule Out Myocardial Infarction using Computer Assisted Tomography (ROMICAT) trial. Am Heart J. 2009 Oct;158(4):562-8. doi: 10.1016/j.ahj.2009.07.027. PMID 19781415
- [Result] Truong QA, Toepker M, Mahabadi AA, Bamberg F, Rogers IS, Blankstein R, Brady TJ, Nagurney JT, Hoffmann U. Relation of left ventricular mass and concentric remodeling to extent of coronary artery disease by computed tomography in patients without left ventricular hypertrophy: ROMICAT study. J Hypertens. 2009 Dec;27(12):2472-82. doi: 10.1097/HJH.0b013e328331054a. PMID 19696685
- [Result] Hoffmann U, Nagurney JT, Moselewski F, Pena A, Ferencik M, Chae CU, Cury RC, Butler J, Abbara S, Brown DF, Manini A, Nichols JH, Achenbach S, Brady TJ. Coronary multidetector computed tomography in the assessment of patients with acute chest pain. Circulation. 2006 Nov 21;114(21):2251-60. doi: 10.1161/CIRCULATIONAHA.106.634808. Epub 2006 Oct 30. PMID 17075011
- [Derived] Karady J, Mayrhofer T, Ferencik M, Nagurney JT, Udelson JE, Kammerlander AA, Fleg JL, Peacock WF, Januzzi JL Jr, Koenig W, Hoffmann U. Discordance of High-Sensitivity Troponin Assays in Patients With Suspected Acute Coronary Syndromes. J Am Coll Cardiol. 2021 Mar 30;77(12):1487-1499. doi: 10.1016/j.jacc.2021.01.046. PMID 33766254
- [Derived] Ferencik M, Mayrhofer T, Lu MT, Woodard PK, Truong QA, Peacock WF, Bamberg F, Sun BC, Fleg JL, Nagurney JT, Udelson JE, Koenig W, Januzzi JL, Hoffmann U. High-Sensitivity Cardiac Troponin I as a Gatekeeper for Coronary Computed Tomography Angiography and Stress Testing in Patients with Acute Chest Pain. Clin Chem. 2017 Nov;63(11):1724-1733. doi: 10.1373/clinchem.2017.275552. Epub 2017 Sep 18. PMID 28923845
- [Derived] Pursnani A, Lee AM, Mayrhofer T, Ahmed W, Uthamalingam S, Ferencik M, Puchner SB, Bamberg F, Schlett CL, Udelson J, Hoffmann U, Ghoshhajra BB. Early resting myocardial computed tomography perfusion for the detection of acute coronary syndrome in patients with coronary artery disease. Circ Cardiovasc Imaging. 2015 Mar;8(3):e002404. doi: 10.1161/CIRCIMAGING.114.002404. PMID 25752898
- [Derived] Hulten E, Goehler A, Bittencourt MS, Bamberg F, Schlett CL, Truong QA, Nichols J, Nasir K, Rogers IS, Gazelle SG, Nagurney JT, Hoffmann U, Blankstein R. Cost and resource utilization associated with use of computed tomography to evaluate chest pain in the emergency department: the Rule Out Myocardial Infarction using Computer Assisted Tomography (ROMICAT) study. Circ Cardiovasc Qual Outcomes. 2013 Sep 1;6(5):514-24. doi: 10.1161/CIRCOUTCOMES.113.000244. Epub 2013 Sep 10. PMID 24021693
- [Derived] Seneviratne SK, Truong QA, Bamberg F, Rogers IS, Shapiro MD, Schlett CL, Chae CU, Cury R, Abbara S, Brady TJ, Nagurney JT, Hoffmann U. Incremental diagnostic value of regional left ventricular function over coronary assessment by cardiac computed tomography for the detection of acute coronary syndrome in patients with acute chest pain: from the ROMICAT trial. Circ Cardiovasc Imaging. 2010 Jul;3(4):375-83. doi: 10.1161/CIRCIMAGING.109.892638. Epub 2010 May 19. PMID 20484542